CLINICAL TRIAL: NCT04483635
Title: PROTECT RCT (PRevention of COVID-19 With Oral Vitamin D Supplemental Therapy in Essential healthCare Teams
Brief Title: PRevention of COVID-19 With Oral Vitamin D Supplemental Therapy in Essential healthCare Teams
Acronym: PROTECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A premature discontinuation was recommended by the Data Safety Monitoring Board and agreed upon by the principal investigator, because the significantly lower recruitment than planned, in the context of mass vaccination of the target population.
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laboratoire RIVA (Unknown)
Responsible Party: Principal Investigator, Professor Francine Ducharme, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MP-21-2021-3044
Record Dates: First submitted 2020-06-29; First posted 2020-07-23 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Vitamin D; Primary prevention; Health care workers
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel-group, placebo controlled trial of vitamin D3 supplementation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Laboratoires Riva will provide the active vitamin D3 and placebo pills, identical in appearance, which will be pre-packaged in coded 60-pill bottles. A web-based randomisation system will allow the research personnel (RP) to log in, obtain a randomization number, and dispense study drugs, pre-prepared by the Central pharmacy, in masked kits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 10 placebo tablets taken orally at baseline, followed by 1 placebo tablet once a week for 16 weeks
  Note that the study may be prolonged according to the overall infection rate monitored monthly.
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 (Experimental): 10 tablets containing 10,000 IU (total : 100,000 IU) of Vitamin D3 taken orally at baseline, followed by 10,000 IU once a week for 16 weeks.
  Note that the study may be prolonged according to the overall infection rate monitored monthly.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Placebo — Weekly oral dose of placebo
  Arms: Placebo
Dietary Supplement: Vitamin D — Weekly oral dose of Vitamin D
  Other Names: cholecalciferol
  Arms: Vitamin D3

SUMMARY:
In this 16-week randomized control study, health care workers will receive a bolus dose followed by a weekly dose of vitamin D or a placebo bolus and weekly dose. This study will test whether high-dose of vitamin D supplementation decreases the incidence of laboratory-confirmed COVID19 infection (primary outcome), reduces illness severity, duration, as well as work absenteeism among health care workers (HCW) in setting at high-risk of contact with COVID-19 cases in high COVID-19 incidence areas.

DETAILED DESCRIPTION:
Design. A 16-week triple-blind, placebo-controlled parallel-group, randomised trial of high-dose vitamin D supplementation compared to placebo in health care workers (HCW).

Subjects: HCW caring for individuals at high-risk of infection (i.e., COVID-suspected or confirmed cases) will be randomly allocated in a 1:1 ratio in variable block size to: Intervention-1 oral loading dose of 100,000 IU vitamin D3 + 10000 IU weekly vitamin D3 or Control-identical placebo loading dose + daily placebo. Follow-up: 2 (randomisation and end-of-study) virtual or in-person visits with weekly reminders, brief health and work-status questionnaire.

Randomisation/allocation concealment: Randomisation will be implemented using a computer-generated random list stratified by regions; health care workers will be allocated (1:1) using permuted block randomisation to enhance concealment.

Sample size: A total of 2414 healthcare workers will provide 80% power to detect a 20% reduction in the risk of laboratory-confirmed COVID-19 infection. Given uncertainties in the infection progression, a Bayesian adaptive design is used where the posterior probability of effectiveness is the basis of inference and decision making, for study continuation or termination.

Procedures. Use of remote or in-person randomisation and/or end-of-study visits and remote documentation of outcomes via electronic communication, mailing of biological samples, and external databases will facilitate enrolment, monitoring, and retention of motivated HCW in this high-intensity trial.

Data analyses: An intention-to-treat analysis will be carried out on all randomized participants. Efficacy and safety analyses will be performed under allocation concealment with unblinding occurring after trial completion and analysis of primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* are aged ≥18 and <70 years old;
* licenced to practice in Quebec;
* working or scheduled to work over the next 16 weeks in a setting at high-risk of contact with COVID-19 infected individuals, particularly (but not only) those involved with aerosol generating medical procedures in hospitals and/or caring for patients in long-term care facilities;
* working in high COVID incidence areas;
* covered by the RAMQ for medical services and hospitalisations;
* has a personal email or phone (to which to send every two weeks a reminder and questionnaire by email or text messages);
* has a fixed address (to which to send the material) in the greater Montreal or surrounding areas.

Exclusion Criteria:

* vitamin D supplementation >400 IU/day or >12,000 IU/month in past 3 months;
* intention to take >400 IU per day during the study period;
* suspected or previously documented COVID-19 infection;
* history of nephrolithiasis, hypercalcemia, hyperphosphatemia, hyperparathyroidism, granulomatosis disease (e.g., tuberculosis, sarcoidosis), renal impairment/failure, or active cancer;
* use of any of the following medications: lithium, teriparatide, or digoxin;
* anticipated prolonged absence from work during the study period (i.e., pregnancy);
* enrolment in a concurrent randomized trial;
* has received a vaccine against COVID-19.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Change in incidence of laboratory-confirmed COVID-19 infection | 16 weeks
  documented by salivary or NP samples obtained clinically for screening or diagnostic purposes throughout the study period, self-obtained salivary samples at endpoint, analysed by RT-qPCR or COVID-19 seroconversion at endpoints

SECONDARY OUTCOMES:
Distribution of disease severity | up to 16 weeks
  5-category ordinal variable [asymptomatic, mild (managed at home); moderate (hospitalisation without supplemental oxygen; severe (oxygen supplementation); critical (mechanical ventilation/death)
Duration of symptoms in COVID-19 positive participants | up to 16 weeks
  For asymptomatic positive COVID-19 participants, symptoms will be recorded in a daily diary up to 14 days. Symptomatic positive COVID-19 participants will record their symptoms in a daily diary up to 48 hours after the resolution of symptoms
Number of participants with COVID-19 positive IgG serology | 16 weeks
  SARS-CoV-2 IgG Diasorin on Liaison XL platform
Number of workday absences due to COVID-19 suspected/confirmed infection | 16 weeks
  Participant-reported; reported by Direction of Human Resource (or for physicians, Direction des services professionnelles) databases
Number of workday absences for any reason | 16 weeks
  Participant-reported; reported by Direction of Human Resource (or for physicians, Direction des services professionnelles) databases
Adverse health events | 16 weeks
  Number and distribution of adverse health events

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, MD, Principal Investigator — St. Justine's Hospital; Cecile Tremblay, MD, Principal Investigator — CHUM
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - CHU Sainte-Justine (CHUSJ), Montreal, Quebec

REFERENCES:
- [Derived] Ducharme FM, Tremblay C, Golchi S, Hosseini B, Longo C, White JH, Coviello D, Quach C, Ste-Marie LG, Platt RW. Prevention of COVID-19 with oral vitamin D supplemental therapy in essential healthcare teams (PROTECT): protocol for a multicentre, triple-blind, randomised, placebo-controlled trial. BMJ Open. 2023 May 25;13(5):e064058. doi: 10.1136/bmjopen-2022-064058. PMID 37230524
- [Derived] Hosseini B, Tremblay CL, Longo C, Glochi S, White JH, Quach C, Ste-Marie LG, Platt RW, Ducharme FM. Oral vitamin D supplemental therapy to attain a desired serum 25-hydroxyvitamin D concentration in essential healthcare teams. Trials. 2022 Dec 16;23(1):1019. doi: 10.1186/s13063-022-06944-z. PMID 36527143